CLINICAL TRIAL: NCT03331354
Title: Assessing the Effect of Distance Learning Vocational Rehabilitation on Employment Outcomes of Veterans With Psychiatric Illness and Histories of Legal Convictions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: D2451-R; RX002451 (Other Grant/Funding Number: VA RR&D)
Record Dates: First submitted 2017-10-31; First posted 2017-11-06 (Actual); Results first posted 2024-06-28 (Actual); Last update posted 2024-06-28 (Actual); Status verified 2024-03

CONDITIONS: Unemployment; Mental Illness; Substance Use Disorder; Legal History
Keywords: employment; distance learning; incarceration
MeSH Terms: conditions — Mental Disorders; Substance-Related Disorders

STUDY DESIGN:
Intervention Model Description: Patients will be randomly assigned to either a distance learning program (COMPASS) or basic vocational services.
Who Masked: Outcomes Assessor
Masking Description: Outcomes assessors will be blinded to conditions
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Self-help resources (Active Comparator): a self-help vocational manual
  Interventions: Other: Basic vocational services
- Compass (Experimental): a distant learning vocational program
  Interventions: Behavioral: Distant vocational learning

INTERVENTIONS:
Behavioral: Distant vocational learning — use of hybrid distance learning to facilitate successful employment outcomes
  Other Names: Compass
  Arms: Compass
Other: Basic vocational services — self-help manual
  Other Names: Basic services
  Arms: Self-help resources

SUMMARY:
64,000 Veterans are released annually from jails and prisons. These Veterans have a weekly unemployment rate of up to 40-55%. However, many are unable to access traditional vocational rehabilitation, not to mention specialized vocational rehabilitation for those with felony histories. Distance learning may be effective in improving access to rehabilitation as well as improving employment outcomes. The Compass system was developed to incorporate both synchronous and asynchronous distance learning to provide effective services. This study will evaluate 150 Veterans with histories of legal convictions and mental illness and/or a substance use disorder. Veterans will be randomly assigned to either a basic vocational resources condition or the the Compass condition. In the basic condition, Veterans will be provided with basic information about where they can access vocational services and a paper version of a vocational reintegration manual, specifically the About Face Vocational Manual. Veterans assigned to the Compass condition will be given access to the online instruction through Videos, live chat features, and tele-health practice interviews with feedback. Veterans will be followed for 6 months. The primary outcomes are employment and interview skills.

DETAILED DESCRIPTION:
At this time, there are over 131,000 Veterans in US prisons and over 50,000 in US jails. When discharged, these Veterans will be forced to cope with high rates of psychosocial and health issues including homelessness, divorce, mental illness, and infectious diseases.

One of the most significant consequences of incarceration is a high rate of unemployment. Evaluations of employment find those with felony histories worked, on average, between 10% and 23% fewer hours than those without felony histories. These negative employment outcomes are caused by a combination of eroded skills, poor social connections, legal restrictions, and stigma.

Though the VA offers a number of vocational rehabilitation and reintegration services, these services are typically not targeted towards Veterans with criminal histories. Also the programs have limitations restricting the range of Veterans that can be served. For example, Veterans living a great distance from a major medical center, rural Veterans, homeless Veterans, and Veterans without transportation may have difficulty accessing services.

To reach the most Veterans, tele-health and distance learning methods must be developed to bring services to the Veterans rather than bring the Veterans to the services. Already well integrated into many educational classrooms, distance learning can be a very effective method of imparting training, skills, and information while mitigating many of the logistical limitations encountered by Veterans with histories of incarceration.

To be successful distance learning should incorporate a number of different best practices. Distance learning should be engaging, avoiding long periods of reading. It should focus on small 'chunks' of information to improve learning and retention. Due to differences in learning, a multiple modality approach is most likely to be successful. Questions, short quizzes, and problem based activities with immediate feedback should be used to keep participants both engaged and to assess progress.

An important aspect to effectively implementing distance learning is to provide blended learning or a hybrid between asynchronous learning, where the participant and teacher are not interacting in real-time, and synchronous learning, where the participant and teacher are interacting directly with each other either in person or across some type of medium. Used effectively, hybrid distance learning can bring a number of positives aspects to the learning environment, including the ability to review information and lessons, practice and role playing, more time to reflect on answers, and less pressure to respond in a group.

Based on effective distance learning principles, the Compass system was developed. Compass builds on a previous pilot online system, the About Face Online System (AFOS), which placed a vocational manual into an online fillable format; however, though Veterans engaged the AFOS, a number of limitations were identified that limited Veterans' enthusiasm, including use of extended reading passages, no direct interaction with a person, and not enough focus on interviews.

Compass uses distance learning best practices including the use of both synchronous and asynchronous learning. The asynchronous components of Compass use video and online content. Veterans are also quizzed at each step of the process on what responses should be given through a multiple choice method. Synchronous components of Compass include tele-health practice interviews, phone coaching sessions, and live-chat features that are used to assist Veterans tailor their information and improving their interview skills.

This study is a four-year project to compare the effectiveness of the Compass system to basic resources. 150 Veterans with legal convictions and mental illness and/or substance use disorders will be followed for six months. Half will receive access to the Compass system and half will receive only basic resources (i.e. a hard copy vocational manual). Outcomes evaluated are employment and interview skills.

The goals of the study are:

1. Compare rates of employment of Compass to those receiving basic resources.
2. Compare improvements in interviewing skills between those receiving an online program to those receiving basic resources.

Hypotheses/expected results

1) Veterans using Compass will have superior rates of employment and improved interviewing skills compared to those receiving basic services.

ELIGIBILITY:
Inclusion Criteria:

* mental illness or substance use disorder
* history of a felony conviction or non-traffic related misdemeanor

Exclusion Criteria:

* cognitive impairment which prohibits active participation in study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 136 (Actual)
Dates: Start 2019-05-01 (Actual); Primary Completion 2022-10-03 (Actual); Study Completion 2023-05-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James P. LePage, PhD, Principal Investigator — VA North Texas Health Care System Dallas VA Medical Center, Dallas, TX
Locations (1):
- VA North Texas Health Care System Dallas VA Medical Center, Dallas, TX, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment occurred between 5/13/2019 and 4/28/2022 (during COVID). Recruitment was initially performed on site at the main hospital in VANTHCS (Dallas) but due to COVID, and with IRB approval, remote consenting was allowed.
Pre-assignment Details: The procedures were to review with the Veteran enrollment criteria (inclusion and exclusion), then consent Veteran. After consent, a detailed history (including confirmation of criteria) was scheduled on a different date. If the Veteran did not, they were withdrawn. Of those consented but withdrawn, 12 had no legal history and 2 had no interest in employment. Additionally, 25 Veterans did not return after consenting for the detailed history. A total of 39 Veterans (28%) were not randomized.
Groups:
- Self-help Resources: Basic vocational services using the About Face Vocational self-help manual: Those receiving the hardcopy manual received a self-guided manual developed and described in previous studies. Briefly, the manual consisted of a series of modules which guide the Veteran through determining their vocational skills, answering interview questions, and addressing their legal and employment histories. Veterans' participation was self-paced. Three weeks after receiving the manual, staff contacted the participants and reviewed and recorded the percentage of the manual completed. To determine employment outcomes, veterans were contacted monthly after enrollment and chart notes reviewed.
- Compass: A distant learning vocational program
  Distant vocational learning: Veterans assigned to COMPASS were given access to the online Compass system with content modeled after the About Face Manual of condition 1. Veterans were assigned a vocational rehabilitation specialist (VRS) whom they were never physically in the same room.
  Compass incorporated both asynchronous and synchronous learning. Asynchronous components, accessible at any time, were videos focused on the concepts of successful job search and handling legal history, as well as the ability to interact with Compass by entering personalized information needed for job search into Compass through fillable fields, similar to the About Face Manual. VRS's were also able review of the information inputted into Compass, making comments directly to the system for the Veteran to review through messages in the system, to suggest better phrasing, more details, etc. Synchronous components were 1) a live chat feature allowing Veterans to ask questions directly to the VRS monitoring the system; 2) telephone coaching where veterans may phone a Hot-Line during office hours to review difficult concepts, discuss progress, discuss upcoming interviews, and problem solve barriers; and 3) practice interviews with feedback via telehealth or phone. To determine employment outcomes, veterans were contacted monthly after enrollment and chart notes reviewed.
Period: Overall Study
Arm/Group | Self-help Resources | Compass
Started | 47 | 50
Completed | 43 | 40
Not Completed | 4 | 10
Not completed — Withdrawal by Subject | 1 | 3
Not completed — Lost to Follow-up | 3 | 3
Not completed — Found employment before initiated active intervention | 0 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Self-help Resources | Compass | Total
Number analyzed (Participants) | 43 | 40 | 83
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.3 (8.1) | 55.3 (8.6) | 56.8 (8.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 4 | 9
  Male | 38 | 36 | 74
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 5 | 7
  Not Hispanic or Latino | 41 | 35 | 76
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 38 | 26 | 64
  White | 5 | 14 | 19
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 43 | 40 | 83
Months of incarceration lifetime [Mean (Standard Deviation); unit: Months] | 67.9 (91.9) | 58.4 (77.2) | 63.8 (84.8)
Substance Use Disorder [Count of Participants; unit: Participants] | 39 | 33 | 72
PTSD [Count of Participants; unit: Participants] | 15 | 19 | 34
Depression Diagnosis [Count of Participants; unit: Participants] | 15 | 17 | 32
Comorbid Substance Use Disorder and Mental Illness [Count of Participants; unit: Participants] | 27 | 24 | 51

OUTCOME MEASURES:

1. Primary Outcome: Competitive Employment Within Six Months of Random Assignment.
Description: Competitive Employment within 6 months of randomization. Competitive employment is defined as a paid position open to anyone, at least at minimum wage, and not a sheltered work position such as the VA's Compensated Work Therapy program. Additionally, day labor type activities were not counted as success.
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Self-help Resources | Compass
Number analyzed (Participants) | 43 | 40
Participants | 15 | 25
Statistical Analysis 1: Comparison: Self-help Resources; Test type: Superiority; p = .016, Chi-squared; Cox Proportional Hazard = 1.87

2. Primary Outcome: Interviewing Skills
Description: Changes in Veterans scores on an interviewing rating form (the Veteran Interview Scale) were compared one month after entry into the study. Scores range from 0 to 30. Higher values are better.
Time Frame: one month
Population: Due to COVID restrictions, not all Veterans could return to the VA to complete the second interview or did not have access to video connection to conduct the interview online.
Measure: Mean (Standard Deviation); unit: Change in raw interview scores
Arm/Group | Self-help Resources | Compass
Number analyzed (Participants) | 34 | 37
Change in raw interview scores | 1.0 (4.6) | 4.4 (5.1)
Statistical Analysis 1: Comparison: Self-help Resources vs Compass; Test type: Superiority; p = .008, ANCOVA; Initial interview scores were used as control in the ANCOVA

3. Secondary Outcome: Change in Job Search Self-Efficacy
Description: Change in job-search efficacy scores were compared between systems at enrollment (point 1) and after 30 days using the systems (point 2). The Job Search Efficacy Scale was used (Cronbach's alpha= .93). Range 10 - 50; higher scores indicate more job search efficacy.
Time Frame: 30 days
Population: The number of participants in this evaluation was lower than number recruited. Participants needed to complete the job-search efficacy scale at the 30 day post group assignment point plus or minus 3 days. However, not all participants provided the data within the time constraints due to onsite restrictions due to COVID-19 and inability to access online data collection systems.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Self-help Resources | Compass
Number analyzed (Participants) | 22 | 28
score on a scale | 1.7 (6.0) | 1.2 (5.7)
Statistical Analysis 1: Comparison: Self-help Resources vs Compass; Test type: Superiority; p = .99, ANCOVA; Change in confidence was evaluated using time one as a covariate
Statistical Analysis 2: Comparison: Self-help Resources vs Compass; Test type: Superiority; p = .99, ANCOVA; Interview scores at enrollment were used as a covariate

4. Post Hoc Outcome: Association Between Percent of COMPASS Completed and Improvement in Interview Skills
Description: The percent of the COMPASS program completed was evaluated to determine its association with improved interview scores.
Time Frame: 30 days
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Percent of program completed
Arm/Group | Self-help Resources | Compass
Number analyzed (Participants) | 34 | 37
Percent of program completed | 48 (41) | 47 (40)
Statistical Analysis 1: Comparison: Compass; This post-hoc analysis was performed on only the COMPASS group to determine the association between percent of the online system completed and change in interview scores; Test type: Other; p < .001, Pearson Correlation

ADVERSE EVENTS:
Time Frame: Adverse events were collected over the six month follow-up period
Arm/Group | Self-help Resources | Compass
All-Cause Mortality (participants affected / at risk) | 0/43 | 0/40
Serious Adverse Events (participants affected / at risk) | 0/43 | 1/40
Other Adverse Events (participants affected / at risk) | 0/43 | 0/40
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Self-help Resources (N=43) | Compass (N=40)
Incarcerated (Social circumstances) | 0 (0) | 1 (1) — Incarcerated while in follow-up

LIMITATIONS AND CAVEATS:
There are several areas of limitations to this study which should be noted. Based on initial goals, an N of 88 was anticipated to be at the lower limit for detecting moderate effect sizes; we fell slightly short but recruitment was adequate for our primary analyses. COVID also created an unusual environment for vocational studies with wild fluctuations in local unemployment rates and an inability to recruit in the community.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2022-10-05): https://cdn.clinicaltrials.gov/large-docs/54/NCT03331354/Prot_SAP_ICF_000.pdf